CLINICAL TRIAL: NCT03734419
Title: Clinical Trials on Prediction of Biological Age Using Saliva Samples of Healthy Population, Based on DNA Methylation Status in ELOVL2 Gene
Brief Title: The Use of Aging Biomarkers in Saliva, Based on DNA Methylation Status in Elovl2 to Predict Biological Age
Status: Withdrawn | Type: Observational
Why Stopped: IRB approval was not obtained for this study.
Sponsor: HKGepitherapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: HKG-Epiaging-104
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: epiaging; biological age; chronological age; DNA methylation; ELOVL2-AS1; ELOVL2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is a big change in our understanding of aging in recent years. Recent researches has revealed clock-like patterns of epigenetic change across in humans. The aging involves a timed epigenetic reprogramming. However, this biological clock which ticks in our DNA is affected by our experience, diet, stress, etc. and it could be changed by experience and life style potentially.

The purpose of this study is to develop and test non-invasive biomarkers based on methylation changes in ELOVL2-AS1 gene in saliva samples using a next generation sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy population

Exclusion Criteria:

* Chronic diseases

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of men and women aged from 18 to 100 years old of different ethnicities living in Kazakhstan.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
The Use of Aging Biomarkers in Saliva, Based on DNA Methylation Status in Elovl2 to Predict Biological Age. | 6 months to 1 year
  We will develop the linear model and a threshold value correlated with chronological age of the individuals participated in the current study. The model will be provided to the researchers:
  Methylation score=(CG1*b1+CG2*b2+ CG3*b3+CGn*n) + e
  CG1 is the methylation value of the first CG b1 is the regression coefficient for the first CG and e equals the intercept. n-is a number of CGs in the model
  We will develop the regression coefficient and intercept as well as the DNA methylation values for each individual for each CG.